CLINICAL TRIAL: NCT01270100
Title: Reducing HIV/AIDS and Drug Abuse Among Heroin Addicts Released From Compulsory Rehabilitation in China
Brief Title: Recovery Management Intervention in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Other Study IDs: DA025385; 1R21DA025385-01 (NIH)
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2010-12

CONDITIONS: Methadone; HIV Infections
MeSH Terms: conditions — HIV Infections

ARMS (1):
- Recovery management intervention (Experimental)
  Interventions: Behavioral: Recovery management

INTERVENTIONS:
Behavioral: Recovery management

SUMMARY:
The purpose of the study is to develop and pilot-test a Recovery Management Intervention (RMI) program for heroin addicts released from compulsory rehabilitation in China.

The project has the following specific aims:

Primary aims:

Aim 1. To engage key stakeholders in the local communities involved in supporting the transition of heroin addicts released from compulsory rehabilitation to the community; Aim 2. To identify potential barriers for participating in MMT in China; Aim 3. To develop and deliver educational/training materials on HIV risks, relapse prevention, and MMT; Aim 4. To adapt and develop the Recovery Management Intervention (RMI) program for heroin addicts released from compulsory rehabilitation in China; Aim 5. To conduct a pilot trial and obtain preliminary outcome data associated with RMI, relative to enhanced standard care.

Secondary aim:

Aim 6. To explore predictors of relapse and HIV/AIDS risk behaviors.

It is hypothesized that the intervention will reduce drug use relapse and the negative consequences associated with relapse, including HIV risk behaviors

ELIGIBILITY:
Inclusion Criteria:The study population will be drawn from all adult patients at participating compulsory rehabilitation facilities who:

1. have been incarcerated for at least one year and would have been eligible for MMT at the time of incarceration,
2. have at least 1 month remaining before release,
3. met the DSM-IV criteria for heroin dependence at the time of incarceration,
4. are willing to enroll in methadone maintenance treatment, and
5. are Shanghai residents who reside in the areas of Shanghai targeted by the study.

Exclusion Criteria: Individuals diagnosed with severe mental illness will not be eligible to participate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

REFERENCES:
- [Derived] Hser YI, Fu L, Wu F, Du J, Zhao M. Pilot trial of a recovery management intervention for heroin addicts released from compulsory rehabilitation in China. J Subst Abuse Treat. 2013 Jan;44(1):78-83. doi: 10.1016/j.jsat.2012.03.009. Epub 2012 Apr 18. PMID 22520276